CLINICAL TRIAL: NCT02592837
Title: Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA) Versus Flexible 19G Endobronchial Ultrasound Transbronchial Needle (Flex 19G EBUS-TBNA) in the Assessment of Mediastinal and Hilar Lymphadenopathy: a Randomised Trial
Brief Title: EBUS-TBNA vs Flex 19G EBUS-TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015LF016B
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Lymphadenopathy; Lung Cancer; Sarcoidosis; Lymphoma
Keywords: Endobronchial ultrasound; EBUS; TBNA; Mediastinal ymphadenopathy; Hilar lymphadenopathy; Lung cancer
MeSH Terms: conditions — Lymphadenopathy; Lung Neoplasms; Sarcoidosis; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flex 19G EBUS-TBNA (Experimental): Mediastinal and hilar lymph node sampling using the flexible 19G EBUS-TBNA needle
  Interventions: Device: Flexible 19G EBUS-TBNA needle
- EBUS-TBNA (Active Comparator): Mediastinal and hilar lymph node sampling using a standard 21G EBUS-TBNA needle
  Interventions: Device: 21G EBUS-TBNA needle

INTERVENTIONS:
Device: Flexible 19G EBUS-TBNA needle
  Arms: Flex 19G EBUS-TBNA
Device: 21G EBUS-TBNA needle
  Arms: EBUS-TBNA

SUMMARY:
Endobronchial ultrasound (EBUS) guided transbronchial needle aspiration (EBUS-TBNA) is an excellent tool for sampling enlarged mediastinal and hilar lymph nodes, but only provides needle aspirate samples which are often adequate for cytological examination only. More advanced histopathological and immunocytopathological assessment of tissue samples, which is particularly important in the diagnosis and staging of cancer, is often not possible with the small cellular samples obtained by EBUS-TBNA. A new transbronchial nodal aspiration needle (the Flex 19G EBUS-TBNA needle) has been developed with a larger needle diameter and more flexibility at the distal end, allowing better access to some lymph nodes stations. This needle can be passed down an EBUS scope and can hypothetically circumvent the deficiencies of EBUS-TBNA highlighted above by providing tissue adequate for histological assessment rather than cytological assessment alone.

This study aims to establish whether the use of the Flex 19G EBUS-TBNA needle can improve the diagnostic yield of EBUS sampling procedures compared to the use of the conventional TBNA needle, thereby allowing more accurate diagnoses and reducing the need repeat procedures or more invasive surgical biopsies, without causing an increase in complication rates. Patients with enlarged mediastinal and hilar lymph nodes referred for EBUS-TBNA will be randomised to have their nodes sampled by either the EBUS-TBNA needle (conventional procedure) or the novel Flex 19G EBUS-TBNA needle. The investigators hope to recruit 250 patients over a 24 month period.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for EBUS-TBNA as part of clinical care
* Lymph nodes larger than 10mm in diameter
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Contraindication to needle biopsy (e.g. coagulopathy, anticoagulation, thrombocytopenia)
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
The difference in quality of diagnostic tissue obtained between the two study arms following 4 separate needle punctures per lymph node | 1 week
  Both specimens (cell pellet and tissue fragments) will be assessed by means of a semiquantitative assessment of material (normal lymph node or lesional tissue) present using the formal scoring system described by Mair.

SECONDARY OUTCOMES:
The difference between the two study arms in the percentage of lymph nodes sampled where enough tissue is obtained for complete immunohistochemical and genetic mutation analysis. | 1 week
The difference in complication rates between the two study arms | 1 month
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with sarcoidosis | 1 week
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with lymphoma | 1 week
The difference in sensitivity for detecting sarcoidosis between the two study arms | 1 week
  Sensitivity = True Positives/(True Positives + False Negatives)
The difference in sensitivity for detecting lymphoma between the two study arms | 1 week
  Sensitivity = True Positives/(True Positives + False Negatives)

CONTACTS AND LOCATIONS:
Overall Officials: Pallav L Shah, MBBS MD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided